CLINICAL TRIAL: NCT01894555
Title: Pharmacogenomics of Antiplatelet Response - II
Brief Title: Pharmacogenomics of Antiplatelet Response - II (PARes-II)
Acronym: PARes-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rehan Qayyum, Assistant Professor of Medicine, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K23HL105897-PARes-II; K23HL105897 (NIH)
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Atherothrombosis
Keywords: Platelet Transcriptome; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Aspirin
MeSH Terms: conditions — Thrombosis; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aspirin (Experimental): Participants treated with aspirin - there is no control group. Participant's baseline will act as their control.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 81 mg daily for 4 weeks

SUMMARY:
This clinical trial is examining the effect of 4-week aspirin therapy on platelet transcriptome in persons at high-risk for myocardial infarction or stroke due to family history of early-onset coronary artery disease.

DETAILED DESCRIPTION:
Platelet aggregation can initiate thrombosis on ulcerated arterial plaques resulting in acute coronary syndrome (ACS). There is large variation in platelet aggregation between individuals. As the genetic message to the cell machinery is conveyed through its transcriptome, we hypothesize that much of the variability in platelet function can be explained by transcriptome changes including differences in gene or isoform expression, altered splicing events, or allele-specific expression. Moreover, aspirin modifies gene expression in several cells, but whether it also affects platelet transcriptome has not yet been studied. Our goal is to characterize the platelet transcriptome and identify genes that are up- or down-regulated after 4-week aspirin therapy. A major strength of our study is that it enrolls individuals from European Americans and African Americans and thus will have the ability to study similarities and differences between the two. The study will produce innovative comparative genomic/platelet phenotype data and will provide a potential pharmacogenomic and diagnostic template for the future discovery of novel antiplatelet regimens to prevent thrombosis-related cardiovascular disease events.

ELIGIBILITY:
Inclusion Criteria:

* Participants from the GeneSTAR cohort
* Unaffected with no overt coronary artery disease or serious vascular event (stroke or peripheral vascular disease diagnosis
* Women who are postmenopausal.
* Women who use a reliable contraceptive method; a reliable contraceptive method will be defined as personal history of tubal ligation, ongoing use of intra-uterine device, or ongoing use of oral contraceptive pills.

Exclusion Criteria:

* Presence of any CAD or stroke, transient ischemic attacks, peripheral arterial disease
* Persons taking aspirin, NSAIDS, or any anti-coagulants who are medically unable to stop them for a two week pre-trial
* A history of allergy to aspirin or clopidogrel
* Weight < 60kg
* Age < 45 and > 75 years of age
* A history of recent or any active bleeding
* Serious or current co-morbidity (AIDS, cancer)
* Pregnant women as determined by urine dipstick pregnancy test
* Any aneurysms on cranial magnetic resonance imaging/magnetic resonance angiography (obtained recently in the GeneSTAR participants)
* Blood pressure above >=159/95mmHg
* History of a gastric or duodenal ulcer, or significant gastrointestinal disease, like regional enteritis
* Mental incompetence to make a decision to participate (developmentally disabled, and persons with diagnosed psychiatric disorders-documented in primary care records).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rehan Qayyum, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- See also: Related Info — http://www.genestarstudy.com/PARes-Study-Aspirn-and-Plavix.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aspirin
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (8.0)
Gender [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Race/Ethnicity, Customized [Number; unit: participants]
  African Americans | 22
  Caucasians | 11

OUTCOME MEASURES:

1. Primary Outcome: Changes in Platelet Transcriptome
Description: Comparison of platelet transcriptome before aspirin therapy with platelet transcriptome after aspirin therapy.
  The expression levels of genes before aspirin therapy was compared with the expression level of the genes after aspirin therapy. The expression levels were measured using the FPKM unit (Fragments Per Kilobase of transcript per Million mapped reads). The gene with the highest difference (pre vs. post) in FPKM is being reported with name in the units area and the actual difference in the number area
Time Frame: 4 weeks
Population: The data were analyzed combining results from two studies (33 from this study and additional 24 individuals from study NCT02234427; total population size = 57) to improve the power to detect a difference. Same results are reported for the two studies. Note that the top most gene (HBG1) with the lowest p-value is being reported.
Measure: Mean (Standard Error); unit: FPKM difference for HBG1 Gene
Arm/Group | Aspirin
Number analyzed (Participants) | 57
FPKM difference for HBG1 Gene | 77.1 (19.8)

ADVERSE EVENTS:
Arm/Group | Aspirin
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No